CLINICAL TRIAL: NCT01005862
Title: A Randomized, Investigator And Subject-Blind, Sponsor-Open, Placebo-Controlled Study To Examine The Effects Of PF-04360365 On ABETA In Patients With Alzheimer's Disease And Healthy Volunteers
Brief Title: Effect of PF-04360365 On ABETA In Patients With Alzheimer's Disease And Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9951011
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease antibody leucine ABeta
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04360365 (Experimental)
  Interventions: Biological: PF-04360365
- Placebo (Placebo Comparator): single dose administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PF-04360365 — 10 mg/kg, single dose administered intravenously
  Arms: PF-04360365
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary goal of this study is to evaluate the effect of PF-04360365 on the clearance of ABETA from the CSF (cerebrospinal fluid) in patients with mild Alzheimer's disease and healthy volunteers. Additionally, the study will assess the pharmacokinetics of PF-04360365, pharmacokinetic and pharmacodynamic relationships in plasma and CSF and the safety and tolerability of single doses of PF-04360365 administered to patients with Alzheimer's disease and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential (age 50 and over for Alzheimer's disease patients; 21-45 for healthy volunteers)
* For patients with Alzheimer's Disease: Diagnosis of probable Alzheimer's disease, consistent with criteria from both National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) and Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* Mini-mental status exam score greater than or equal to 20
* Rosen-Modified Hachinski Ischemia Score of < or = 4
* On stable dose of background cholinesterase inhibitor or memantine at least 3 months prior to enrollment

Exclusion Criteria:

* Diagnosis or history of other demential or neurodegenerative disorders
* Diagnosis or history of clinically significant cerebrovascular disease
* Specific findings on magnetic resonance imaging (MRI); cortical infarct, micro hemorrhage, multiple white matter lacunes, extensive white matter abnormalities
* History of autoimmune disorders
* History of allergic or anaphylactic reactions

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fractional Clearance rate of ABeta peptide in CSF | 36 hours

SECONDARY OUTCOMES:
Area under the ratio of CSF labeled/unlabeled ABETA time curve from onset of clearance to 36h following start of infusion | 36 hours
PF-04360365 concentrations and ABETA concentrations in plasma and CSF | 36 hours
Ratio of labeled/unlabeled leucine in plasma and CSF post labeled leucine administration | 36 hours
Adverse events, vital signs, clinical labs, electrocardiograms, physical / neurologic examinations, Columbia Suicide Severity Rating Scale, MRI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, St Louis, Missouri
- Pfizer Investigational Site, Stockholm, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951011&StudyName=Effect%20of%20PF-04360365%20On%20ABETA%20In%20Patients%20With%20Alzheimer%27s%20Disease%20And%20Healthy%20Volunteers